CLINICAL TRIAL: NCT01995344
Title: A Randomised Phase II Study in Metastatic Melanoma to Evaluate the Efficacy of Adoptive Cellular Therapy With Tumour Infiltrating Lymphocytes (TIL) and Assessment of High Versus Low Dose Interleukin-2
Brief Title: TIL Therapy in Metastatic Melanoma and IL2 Dose Assessment
Acronym: METILDA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Christiesponsoredresearch, Professor in Medical Oncology, The Christie NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11_DOG14_12; 2013-001071-20 (EudraCT Number)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; fludarabine; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A: High Dose Interleukin-2 (HD IL2) (Active Comparator): Eligible participants will undergo surgical tumour excision from which TIL will be derived, cultured and expanded. Participants will receive preconditioning chemotherapy with cyclophosphamide (60mg/kg) day -7 and day -6, followed by fludarabine (25mg/m2) day -5 to day -1. The autologous TILs will be re-infused on day 0 and the patients will receive up to 12 doses of intravenous HD IL2
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Genetic: Tumour Infiltrating Lymphocytes; Drug: Interleukin-2
- ARM B: Low Dose Interleukin-2 (LD IL2) (Active Comparator): Eligible participants will undergo surgical tumour excision from which TIL will be derived, cultured and expanded. Participants will receive preconditioning chemotherapy with cyclophosphamide (60mg/kg) day -7 and day -6, followed by fludarabine (25mg/m2) day -5 to day -1. The autologous TILs will be re-infused on day 0 and the patients will receive up to 12 doses of intravenous LD-IL2
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Genetic: Tumour Infiltrating Lymphocytes; Drug: Interleukin-2

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Fludarabine
Genetic: Tumour Infiltrating Lymphocytes
  Other Names: TIL
Drug: Interleukin-2
  Other Names: IL2

SUMMARY:
This is a two arm, open-labelled phase II randomised trial of Tumour Infiltrating Lymphocytes (TIL) in metastatic melanoma patients given with preconditioning chemotherapy and Interleukin-2 (IL2). Eligible patients will undergo surgical tumour excision from which TIL will be derived, cultured and expanded. Patients will receive preconditioning chemotherapy with cyclophosphamide (60mg/kg) day -7 and day -6, followed by fludarabine (25mg/m2) day -5 to day -1. The autologous TILs will be re-infused on day 0 and the patients will receive up to 12 doses of intravenous High Dose Interleukin-2 (HD-IL2) or Low Dose Interleukin-2 (LD-IL2) depending on the randomised arm.

The primary objectives are response rate assessed and compared by CT scans carried out at week 6, week 12 and at 12 weekly intervals thereafter and the evaluation of feasibility and tolerability of TIL therapy with HD-IL2 versus LD-IL2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignant melanoma with confirmed evidence of progressive metastatic disease and to have failed / refused standard therapies.
* They must have resectable metastatic lesion(s) of at least 2cm in diameter.
* There must be measurable / evaluable disease after the surgical resection.
* Patients may have had any previous systemic therapies including anti-CTLA4 (Ipilimumab) agent provided they are otherwise fit for treatment.
* Tumour samples may be taken prior to other systemic therapy if patients wish to store the sample for possible future use.
* Age equal to or greater than 18 years.
* World Health Organisation (WHO) performance status of 0 or 1.
* Life expectancy >3months.
* LVEF > 50% as measured by ECHO/MUGA and satisfactory stress ECHO (if over 60 or had previous cardiotoxic therapy).
* Haemoglobin (Hb) ≥ 9.0 g/dL
* Neutrophils ≥ 1.0 x 109/L
* Platelets (Plts) ≥ 100 x 109/L
* serum bilirubin ≤ 1.5 x ULN
* alanine aminotransferase (ALT) ≤ 5 x ULN
* aspartate aminotransferase (AST) ≤ 5 x ULN
* alkaline phosphatase (ALP) ≤ 5 x ULN
* Serum creatinine ≤ 0.15 mmol/L
* Female patients of child-bearing potential must have a negative serum or urine pregnancy test prior treatment and agree to use appropriate medically approved contraceptive precautions for four weeks prior to entering the trial, during the trial and for six months afterwards.
* Male patients must agree to use barrier method contraception during the TIL treatment and for six months afterwards.
* Full written informed consent

Exclusion Criteria:

* Those receiving radiotherapy, targeted therapy, immunotherapy, systemic steroids, or chemotherapy during the previous four weeks (six weeks for nitrosoureas and Mitomycin-C) prior to treatment or during the course of the treatment.
* All toxic manifestations of previous treatment must have resolved. Exceptions to this are alopecia or certain Grade 1 toxicities, which an investigator considers should not exclude the patient.
* Previous radiotherapy treatment to the resectable metastatic site(s) within 1 year and no other suitable metastatic sites.
* Participation in any other clinical trial within the previous 30 days or during the course of this treatment.
* Previous allogeneic transplant.
* Patient with ocular melanoma.
* Clinically significant cardiac disease. Examples would include unstable coronary artery disease, myocardial infarction within 6 months or Class III or IV AHA criteria for heart disease (see Appendix 6)
* Patients who are high medical risks because of non-malignant systemic disease, including those with, uncontrolled cardiac or respiratory disease, or other serious medical or psychiatric disorders which in the lead clinicians opinion would not make the patient a good candidate for this therapy.
* Concurrent systemic infections (CTCAE Grade 3 or more) within the 28 days prior to treatment.
* Prior history of malignancies at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin.
* Patients known or found to be serologically positive for Hepatitis B, C, HIV or HTLV.
* History of systemic autoimmune disease which could be life-threatening if reactivation occurred (for example hypothyroidism would be permissible, prior rheumatoid arthritis or SLE would not).
* Patients with more than 3 brain metastases.
* Patients with symptomatic brain metastasis measuring more than 10mm in diameter or evidence of significant surrounding oedema on MRI will not be eligible until after treatment demonstrating no clinical or radiologic CNS progression for at least 2 months. Patient must be able to wean off any steroid use 3 weeks before treatment commencement.
* Patients who are likely to require long-term systemic steroids or other immunosuppressive therapy.
* Pregnant and lactating women.
* Radiotherapy to >25% skeleton.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03-01; Primary Completion 2015-07-24 (Actual); Study Completion 2015-07-24 (Actual)

PRIMARY OUTCOMES:
Disease response according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Best response
  Subject will have CT scan at 6,12,24 weeks post treatment to compare with baseline CT scan in order to assess disease response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul Lorigan, MD, Principal Investigator — The Christie NHS Foundation Trust; Robert E Hawkins, MD, Principal Investigator — The University of Manchester
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom